CLINICAL TRIAL: NCT02874274
Title: Vaccination Uptake in Parkinson's Disease
Brief Title: Vaccination Uptake (VAX) in PD
Acronym: VAX-PD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 16-01157
Record Dates: First submitted 2016-08-17; First posted 2016-08-22 (Estimated); Last update posted 2020-01-10 (Actual); Status verified 2020-01

CONDITIONS: Parkinson's Disease
Keywords: Corticobasal syndrome; Dementia with Lewy Bodies; Home Visit Program (HVP); Multidimensional Caregiver Strain Index; Parkinson's Disease Dementia; Progressive Supranuclear Palsy
MeSH Terms: conditions — Parkinson Disease; Corticobasal Degeneration; Lewy Body Disease; Supranuclear Palsy, Progressive | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- 100 Non-Homebound Subjects (Active Comparator): outpatient healthcare utilization and self-reported illness.
  Interventions: Behavioral: Standard of Care
- 60 Homebound Subjects (Active Comparator): Will test the feasibility of offering influenza and pneumococcal vaccinations, as appropriate, to the homebound individuals in our HVP cohort
  Interventions: Behavioral: Home Visit Program (HVP)

INTERVENTIONS:
Behavioral: Standard of Care
  Arms: 100 Non-Homebound Subjects
Behavioral: Home Visit Program (HVP) — The study team will also contact the subject by phone within one week of each vaccination visit to assess for any adverse effects related to vaccination, included but not limited to: injection site pain, tenderness, swelling, pruritus, induration, or erythema; systemic symptoms such as fatigue, chills, headache, anorexia, malaise, myalgias, or anaphylaxis. Subjects will be contacted 90 days (+ 14 days) following Visit 3 to inquire about any additional symptoms and healthcare utilization.
  Arms: 60 Homebound Subjects

SUMMARY:
This is a study to see whether participation in the Edmond J. Safra Interdisciplinary Home Visit Program for Advanced Parkinson's (HVP) increases the rate of age-appropriate vaccinations in people with advanced Parkinson's Disease (PD) and related disorders. This study will evaluate the impact of the HVP on the rate of common illnesses such as flu and pneumonia in patients with advanced PD and related disorders over the course of one year.

As there is currently no data available on the baseline rate of vaccinations in either homebound or less disabled PD populations, investigators will seek to establish the baseline rate of vaccinations, barriers to getting vaccinated, and baseline healthcare utilization in these populations by piloting (Phase 1) and then implementing (Phase 2) a survey via telephone interviews. Investigators will then test feasibility of offering influenza and pneumococcal vaccinations, as appropriate, to the homebound individuals in our HVP cohort (Phase 3), and will compare their pre- and post-intervention rates of both outpatient and acute healthcare utilization and self-reported illness.

ELIGIBILITY:
Inclusion Criteria:

Phase 1:

* Diagnosed with idiopathic Parkinson's disease (a chronic, slowly-progressive neurological disorder), or related disorders including Dementia with Lewy Bodies, Multiple System Atrophy, Progressive Supranuclear Palsy, or Corticobasal Syndrome.

Phase 2:

* Subjects will be those diagnosed with idiopathic Parkinson's disease (a chronic, slowly-progressive neurological disorder), or related disorders including Dementia with Lewy Bodies, Multiple System Atrophy, Progressive Supranuclear Palsy, or Corticobasal Syndrome.
* Each subject must either 1) be willing and able to provide verbal, informed consent for the study, and for whom capacity to consent will be assessed using the questions below, or 2) if unable to provide informed consent due to lack of capacity, a caregiver is able to provide informed consent and the subject provides assent to participation.

Phase 3:

* Diagnosed with idiopathic Parkinson's disease (a chronic, slowly-progressive neurological disorder), or related disorders including Dementia with Lewy Bodies, Multiple System Atrophy, Progressive Supranuclear Palsy, or Corticobasal Syndrome.
* Each subject must either 1) be willing and able to provide written, informed consent for the study, and for whom capacity to consent will be assessed using the questions below, or 2) if unable to provide informed consent due to lack of capacity, a caregiver is able to provide informed consent and the subject provides assent to participation.

Subjects have one or more of the following criteria:

* Fluctuation
* Multi-morbidity
* Mismanages medication
* Cognitive impairment
* High risk for re-hospitalization
* High risk for nursing facility admission
* Suspected elder abuse
* Recent history of increased falls in home
* Caregiver burnout suspected
* Ability to participate in the research study as deemed by the Principal Investigator.

Exclusion Criteria:

* Diagnosis of another neurodegenerative disease or other major central nervous system disorder.

Subjects with severe hearing impairment or speech dysfunction that would preclude pa -Subjects with active psychosis or exhibiting symptoms of a severe psychiatric disorder.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 164 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2018-04-12 (Actual); Study Completion 2018-04-12 (Actual)

PRIMARY OUTCOMES:
Unified Parkinson's Disease Rating Scale (UPDRS) | 30 Minutes
  A rating scale used to follow the longitudinal course of Parkinson's disease
Hoehn and Yahr Scale (HY) | 30 Minutes
  A system used for describing how Parkinson's symptoms progress and the relative level of disability. There are five stages: Stage 0 - No signs of disease; Stage 1 - Unilateral disease; Stage 1.5 - Unilateral plus axial involvement; Stage 2 - Bilateral disease, without impairment of balance; Stage 2.5 - Mild bilateral disease with recovery on pull test; Stage 3 - Mild to moderate bilateral disease; some postural instability; physically independent; Stage 4 - Severe disability; still able to walk or stand unassisted; Stage 5 - Wheelchair bound or bedridden unless aided.
Parkinson's Disease Questionnaire- Short Form (PDQ-8 | 30 Minutes
  A validated, brief, 8-item measure of quality of life in PD with a summary index score standardized to a scale of 0-100, with higher scores signifying worse quality of life; this scale is recommended for use in PD by the Movement Disorder Society.10

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Feigin, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States